CLINICAL TRIAL: NCT00917657
Title: Corneal Wavefront-Guided PRK With Adjunctive Mitomycin-C for the Treatment of Hyperopia After Radial Keratotomy
Brief Title: Photorefractive Keratectomy (PRK) for Hyperopia After Radial Keratotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Prof. Newton Kara-José, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1183/07
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Hyperopia
Keywords: photorefractive keratectomy; hyperopia; radial keratotomy; refractive surgery
MeSH Terms: conditions — Hyperopia | interventions — Photorefractive Keratectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Photorefractive keratectomy

SUMMARY:
To assess the efficacy, predictability, stability and safety of corneal wavefront-guided photorefractive keratectomy (PRK) for correcting hyperopia and astigmatism after radial keratotomy (RK).

ELIGIBILITY:
Inclusion Criteria:

* Hyperopia or hyperopic astigmatism with spherical equivalent of up to + 9,25 D and astigmatism of up to - 4,5 D;
* Uncorrected Visual Acuity of 20/40 or worse;
* Best-Corrected Visual Acuity of 20/60 or better.

Exclusion Criteria:

* Systemic or ocular conditions that could bias results
* Previous photorefractive surgery

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

REFERENCES:
- [Derived] Ghanem RC, Ghanem EA, Kara-Jose N. [Safety of photorefractive keratectomy with mitomycin-C for the treatment of hyperopia after radial keratotomy]. Arq Bras Oftalmol. 2010 Mar-Apr;73(2):165-70. doi: 10.1590/s0004-27492010000200013. Portuguese. PMID 20549047
- [Derived] Ghanem RC, Ghanem EA, Kara-Jose N. [Corneal wavefront-guided photorefractive keratectomy with mitomycin-C for consecutive hyperopia after radial keratotomy]. Arq Bras Oftalmol. 2010 Jan-Feb;73(1):70-6. doi: 10.1590/s0004-27492010000100013. Portuguese. PMID 20464118